CLINICAL TRIAL: NCT06507449
Title: The Influence of Modifying Highly Calcified Coronary Lesions on Coronary Microcirculation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Polish Cardiac Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BNW/NWN/0052/KB1/4/24
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Calcification; Ischemic Heart Disease; Non-ST-Segment Elevation Myocardial Infarction (NSTEMI); Coronary Artery Disease; Angina, Unstable; Tomography, Optical Coherence
Keywords: Percutaneous coronary intervention; Microcirculation
MeSH Terms: conditions — Myocardial Ischemia; Non-ST Elevated Myocardial Infarction; Coronary Artery Disease; Angina, Unstable | interventions — Lithotripsy; Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- High-pressure non-compliant balloon (Experimental): The SIS Medical OPN NC® super high-pressure coronary balloon will be used for balloon angioplasty vessel preparation prior to implantation of a drug-eluting stent.
  Interventions: Device: High-pressure non-compliant balloon; Device: Optical coherence tomography; Device: Coroventis Coroflow Cardiovascular System and PressureWire™ X Guidewire
- Orbital atherectomy (Experimental): The Diamondback 360® Coronary Orbital Atherectomy System (OAS) will be used for orbital atherectomy (OA) vessel preparation prior to implantation of a drug-eluting stent.
  Interventions: Device: Orbital atherectomy; Device: Optical coherence tomography; Device: Coroventis Coroflow Cardiovascular System and PressureWire™ X Guidewire
- Lithotripsy (Experimental): The Shockwave® Medical system will be used for intravascular lithotripsy (IVL) vessel preparation prior to implantation of a drug-eluting stent.
  Interventions: Device: Lithotripsy; Device: Optical coherence tomography; Device: Coroventis Coroflow Cardiovascular System and PressureWire™ X Guidewire

INTERVENTIONS:
Device: Lithotripsy — Calcified lesion preparation using lithotripsy before implantation of a drug-eluting stent
  Arms: Lithotripsy
Device: Orbital atherectomy — Calcified lesion preparation using orbital atherectomy before implantation of a drug-eluting stent
  Arms: Orbital atherectomy
Device: High-pressure non-compliant balloon — Calcified lesion preparation using high-pressure non-compliant balloon before implantation of a drug-eluting stent
  Arms: High-pressure non-compliant balloon
Device: Optical coherence tomography — Optical coherence tomography assessment of coronary arteries.
Device: Coroventis Coroflow Cardiovascular System and PressureWire™ X Guidewire — A coronary thermodilution system used for evaluate differences between the impact of calcified lesion preparation methods on coronary microvascular function.

SUMMARY:
This is a prospective, single-center, three-arm study to evaluate the impact of severely calcified coronary lesions treatment on microvascular circulation. We will enroll 30 conveniently sampled subjects assigned to one of three therapeutical methods lithotripsy, super-high pressure balloon, and orbital atherectomy prior to implantation of drug-eluting stents (DES).

DETAILED DESCRIPTION:
This prospective, non-randomized, single-center study includes subjects who meet all of the inclusion and none of the exclusion criteria and sign the ICF. 30 patients with severe coronary stenosis will be enrolled. The severity will be assessed by Optical Coherence Tomography (OCT) based on the degree of calcification in the coronary lesion as defined by this protocol. Subjects will be assigned to one of three arms (lithotripsy, super-high pressure balloon or orbital atherectomy) followed by an implantation of drug-eluting stents (DES). The aposition and expansion of DES will be evaluated using OCT . Patients will be followed through discharge, 30 days and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with native coronary artery disease (including stable or unstable angina and NSTEMI) suitable for PCI.
* The lesion must be crossable with the study guide wire.
* The target vessel reference diameter must be ≥ 2.5mm and ≤ 4.0 mm.
* The target lesion must have evidence of severe calcium deposit at the lesion site based on the protocol criterion.
* Subject or legally authorized representative, signs a written Informed Consent form to participate in the study, prior to any study-mandated procedures.
* Male or female, age above or equal to 18 years at the time of signing informed consent.

Further inclusion criteria may apply

Exclusion Criteria:

* Inability to understand the study or a history of non-compliance with medical advice.
* Unwilling or unable to sign the Informed Consent Form (ICF).
* History of any cognitive or mental health status that would interfere with trial participation.
* Male or female, age under 18 years at the time of signing informed consent.
* Female subjects who are pregnant or planning to become pregnant within the study period.
* Subject has a known sensitivity to contrast media, which cannot be adequately pre-medicated.
* Subject has evidence of an active infection on the day of the procedure requiring oral or intravenous antibiotics.
* Limited long term prognosis due to other conditions.
* Subjects in cardiogenic shock or with decompensated heart failure (NYHA class IV).
* Subject diagnosed with chronic kidney disease stage 4 or greater (eGFR <30).
* Most recent left ventricular ejection fraction ≤ 20%.
* Subject is an acceptable candidate for coronary artery bypass surgery.
* The target vessel reference diameter is under 2.0 mm.
* Target lesion is located in or supplied by an arterial or venous bypass graft.
* The target vessel has angiographically visible or suspected thrombus.
* The target lesion is in an in-stent restenosis.
* Subject has received a heart transplant.
* Subject has major valve disease and underwent intervention within 30 days prior to randomization.

Further exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Coronary Flow Reserve (CFR) | Intraprocedural
  Determination of a difference between Coronary Flow Reserve (CFR) at the beginning and at the end of the procedure using CoroFlow™ Cardiovascular System.
Index of Microcirculatory Resistance (IMR) | Intraprocedural
  Determination of a difference between Index of Microcirculatory Resistance (IMR) at the beginning and at the end of the procedure using CoroFlow™ Cardiovascular System.

SECONDARY OUTCOMES:
Stent expansion | Intraprocedural
  Stent expansion (%) evaluated by optical coherence tomography.
Acceptable stent expansion | Intraprocedural
  Acceptable stent expansion (cut-off value defined as >80%) evaluated by optical coherence tomography.
Optimal stent expansion | Intraprocedural
  Optimal stent expansion (cut-off value defined as >90%) evaluated by optical coherence tomography.
Minimal lumen diameter (MLD) difference | Intraprocedural
  Determination of a difference between quantitative OCT measured minimal lumen diameter (MLD) at the beginning and at the end of the procedure.
Procedural Success | Up to 3 years
  Procedural success - defined as successful stent delivery and angiographic in-vessel residual stenosis <30%, and with the absence of any of the following: stent loss, coronary artery dissection, coronary artery perforation, PCI no reflow phenomenon or MACCE (defined as a composite of cardiovascular death, myocardial infarction at the targeted vessel, targeted coronary vessel revascularization (PCI or CABG), TIA or stroke).
Strategy Success | Intraprocedural
  Strategy success - defined as procedural success without crossover to alternative treatment.

OTHER OUTCOMES:
The proportion of subjects that experience Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | Up to 3 years
  30-day and 1 year MACCE defined as a composite of cardiovascular death, myocardial infarction at the targeted vessel, targeted coronary vessel revascularization (PCI or CABG), TIA or stroke.
The proportion of subjects that experience Target Vessel Revascularization (TVR) | Up to 3 years
  30-day and 1 year Target Vessel Revascularization (TVR) - defined as any repeat revascularization at the target vessel (inclusive of the target lesion) and target vessel collaterals after the completion of the procedure.
The proportion of subjects that experience Target Lesion Revascularization (TLR) | Up to 3 years
  30-day and 1 year Target Lesion Revascularization (TLR) - defined as repeat intervention PCI or surgery within the index procedure stent or 5mm proximal or distal to the stent.
Myocardial infarction (MI) rate at 30-day and 1 year | Up to 3 years
  The proportion of subjects that experience a Myocardial Infarction (MI) at 30-day and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Gąsior, MD, PhD, Principal Investigator — Division of Cardiology and Structural Heart Diseases, Medical University of Silesia
Locations (1):
- Upper Silesian Medical Centre, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No